CLINICAL TRIAL: NCT00209508
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 2-Year Study To Evaluate The Effects Of GPI 1485 On [123I]b-CIT/SPECT Scanning And Clinical Efficacy In Symptomatic PD Patients Receiving Dopamine Agonist Therapy.
Brief Title: 2 Year Study to Evaluate the Effects of GPI 1485 on [123I]b-CIT/SPECTScanning and Clinical Efficacy in Patients With PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Symphony Neuro Development Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0501-0201
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; SPECT Scanning
MeSH Terms: conditions — Parkinson Disease | interventions — GPI 1485

INTERVENTIONS:
Drug: GPI 1485

SUMMARY:
This study was designed to assess whether GPI 1485 has the ability to delay or stop disease progression and improve symptoms in patients with Parkinson's disease (PD) that is already being treated with a dopamine agonist therapy. Whether the drug is working will be assessed by evaluating clinical endpoints such as UPDRS scores and by evaluating images, obtained by SPECT scan, of brain activity. Participants in the study will be given either placebo or GPI 1485 treatment. The duration of the study is 2-years and patients are required to complete 12 safety visits and 3 SPECT scans. SPECT scans will be taken before, after 1-year, and after 2-years of treatment with GPI 1485. In completing the SPECT scan, patients will be injected with a radioactive investigational drug b-CIT and pictures taken using a Single Photon Emission Computed Tomography (SPECT) camera.

DETAILED DESCRIPTION:
In this phase II study, the investigational new drug (not approved by the FDA) GPI 1485 is being assessed for its ability to delay or stop disease progression and improve symptoms in patients with mild to moderate Parkinson's disease (PD). These potential effects of GPI 1485 are based on animal studies in which the drug was shown to both protect nerves from damage and to regrow damaged nerves. Participants in this study will be randomly assigned to receive either GPI 1485 or placebo (inactive pill). GPI 1485 will be supplied as an oral tablet formulation to participants enrolled in the study. Participants randomly assigned to receive GPI 1485 will be required to take four tablets four times a day by mouth. GPI 1485 matching placebo will also be supplied as an oral tablet formulation. Participants randomly assigned to placebo will be required to take four placebo tablets four times a day by mouth. The duration of this study is 24 months which includes 12 clinical visits at one of 21 participating sites and three imaging visits to Molecular NeuroImaging (MNI) in New Haven Connecticut. At MNI, participants will be injected with a radioactive investigational drug b-CIT to obtain images of the activity in the brain with Single Photon Emission Computed Tomography (SPECT). This will evaluate whether GPI 1485 slows or delays the loss of brain activity in patients with mild to moderate PD. During this study you will also have other clinical evaluations including a physical exam, blood work, ECG (tracing of your heart rhythm), and urinalysis. Tests specific to Parkinson's disease will also be performed including: Unified Parkinson's Disease Rating Scale (UPDRS), Dyskinesia Rating Scale, Bilateral finger-tapping test, and Parkinson's Disease Sleep Scale (PDSS). In addition assessments of your health and mood will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 40 - 80 years of age with a diagnosis of idiopathic PD < 10 years. The diagnosis of idiopathic PD will be based on the medical history, neurologic examination, current response to anti-PD medication(s), and the presence of at least two of the following at the time of diagnosis: resting tremor, bradykinesia, or rigidity.
2. Females must be postmenopausal for >= 12 months, surgically sterile, or agree to use acceptable forms of contraception. A negative serum pregnancy test must be confirmed prior to first dose for women of childbearing potential.
3. Clinical diagnosis of idiopathic mild to moderate PD characterized by a Hoehn and Yahr rating of 1 to 3 in the 'Off' state (measured before the first dose of anti-PD medications on the day of assessment).
4. UPDRS Motor 'Off' rating of 8-30 (measured before the first dose of anti-PD medications on the day of assessment).
5. Mini-Mental Status Examination (MMSE) score of <= 25.
6. Currently treated with an optimized dose of a dopamine agonist (stable dose for >= 1 month prior to randomization and treatment is optimized in the opinion of the Investigator).
7. In the judgment of the Investigator the patient will not require L-Dopa therapy within the 3 months after randomization.
8. Concomitant therapy with amantadine, selegiline, or anticholinergics is permitted, but not required. If the patient is treated with any of these medications the dose of this medication must be judged optimal and stable for > 1 month prior to randomization.

Exclusion Criteria:

1. Presence of motor fluctuations including drug-induced dyskinesia, but excluding the pre-dose 'Off' state (prior to the first dose of anti-parkinsonian medication(s) on the day of assessment).
2. History of surgical treatment of PD.
3. Presence of clinical signs consistent with a neurologic disorder other than PD including, but not limited to, progressive supranuclear palsy, multiple system atrophy (Shy-Drager syndrome, olivopontocerebellar degeneration, striatonigral degeneration), corticobasal degeneration, Pick's disease, diffuse Lewy body disease, dementia, schizophrenia, psychosis, or hallucinations.
4. Presence of clinically significant depression as measured by the HAM-D Scale with a score > 16. If the patient is on an antidepressant, the dose must be judged optimal and stable for ³ 1 month prior to randomization.
5. Presence of clinically significant, in the judgment of the Investigator, urinary incontinence, cardiac arrhythmia, or symptomatic orthostatic hypotension.
6. History of seizure disorder or the occurrence of 1 or more seizures within 1 year before screening.
7. Any medical disability (e.g., peptic ulcer disease, severe degenerative arthritis, compromised nutritional state) or laboratory abnormality (e.g., serum creatinine > 2.0 mg/dL) that may interfere with the protocol-specified safety and efficacy measurements, present an unacceptable risk to the patient's well-being, or compromise the patient's ability to provide informed consent.
8. Recent history, within the 2 years before screening, of drug or alcohol abuse.
9. History of anaphylaxis.
10. Previous treatment with L-Dopa for > 90 days or treatment with L-Dopa within 30 days prior to the baseline assessment.
11. Treatment within the 3 months before the Baseline SPECT Scan with modafinil.
12. Treatment within the 6 months before screening with neuroleptics, methylphenidate, metoclopramide, cinnarizine, flunarizine, reserpine, alpha methyldopa, amphetamine, or monoamine oxidase-A (MOA-A) inhibitors.
13. Previous exposure to GPI 1485 (previously AMG-474-00).
14. Treatment with an investigational agent within the 30 days before screening or scheduled to receive an investigational agent other than that specified by this protocol during the course of this study.
15. Females that are pregnant, breast feeding, or do not agree to use an acceptable form of contraception.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-11; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of GPI 1485 vs. placebo on the percent change from baseline in [123I]ß-CIT/SPECT striatal uptake over 2 years in patients with idiopathic PD.

SECONDARY OUTCOMES:
To evaluate the efficacy of GPI 1485 vs. placebo in the treatment of symptomatic idiopathic PD patients using the following prespecified clinical measures of greatest interest:
Mean daily L-Dopa Therapy Equivalents
UPDRS ('On')
Measures of sleep
Cognitive function
To evaluate the efficacy of GPI 1485 versus placebo using the following other acceptable measures of clinical assessment.
To evaluate the efficacy of GPI 1485 versus placebo on the percent change from baseline in [123I]ß-CIT/SPECT putamen and caudate uptake over 2 years in patients with idiopathic PD.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Favit-Van Pelt, MD, PhD, Study Director — Eisai Inc.